CLINICAL TRIAL: NCT03238924
Title: Augmenting Prolonged Exposure Therapy for PTSD With Intranasal Oxytocin
Brief Title: Prolonged Exposure and Oxytocin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Julianne Flanagan, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 36616
Record Dates: First submitted 2017-04-03; First posted 2017-08-03 (Actual); Results first posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-04

CONDITIONS: PTSD
Keywords: posttraumatic stress disorder; oxytocin; Prolonged Exposure
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): 40 IU intranasal oxytocin spray
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo is matching saline nasal spray
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Oxytocin — 40 IU oxytocin nasal spray, self-administered
  Other Names: Pitocin
  Arms: Oxytocin
Drug: Placebos — Saline nasal spray, self-administered
  Arms: Placebo

SUMMARY:
Posttraumatic stress disorder (PTSD) is a chronic, debilitating anxiety disorder that may develop after direct or indirect exposure to traumatic events. Prolonged Exposure (PE) is a cognitive-behavioral psychotherapy modality with a wealth of empirical support demonstrating its efficacy to treat PTSD in a variety of populations. The neuropeptide oxytocin is a promising new pharmacotherapeutic agent with prominent anxiolytic effects . Despite a strong biological and theoretical rationale for investigating the potential effectiveness of augmenting PE with intranasal oxytocin, no studies to date have done so. The current study aims to address this important gap in the literature by examining changes in PTSD symptoms following PE treatment combined with a) 40 IU of intranasal oxytocin or b) placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; any race or ethnicity; age 18-75 years.
2. Able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of the assessment instruments.
3. Participants must be able to comprehend English.
4. Meet DSM-5 criteria for current PTSD (assessed via the Clinician Administered PTSD Scale; CAPS).
5. A CAPS score of 50 or greater.
6. Participants may also meet criteria for a mood disorder (except bipolar affective disorder, see Exclusion Criteria) or anxiety disorders (e.g., agoraphobia, social phobia, generalized anxiety disorder). The inclusion of participants with affective and anxiety disorders is essential because of the marked frequency of the co-existence of mood and other anxiety disorders among patients with PTSD.
7. Participants taking psychotropic medications will be required to be maintained on a stable dose for at least eight weeks before study initiation. Initiation or change of psychotropic medications during the course of the trial may interfere with interpretation of results.

Exclusion Criteria:

1. Participants meeting DSM-5 criteria for a history of or current psychotic or bipolar affective disorders, or with current suicidal or homicidal ideation and intent. Those participants will be referred clinically.
2. Participants who would present a serious suicide risk or who are likely to require hospitalization during the course of the study. Those participants will be referred clinically.
3. Participants on maintenance anxiolytic, antidepressant, or mood stabilizing medications, which have been initiated during the past 8 weeks.
4. Participants meeting DSM-5 criteria for a substance use disorder, except caffeine or nicotine, within the past 12 months.
5. Pregnant women will be excluded from the proposed study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flanagan JC, Sippel LM, Wahlquist A, Moran-Santa Maria MM, Back SE. Augmenting Prolonged Exposure therapy for PTSD with intranasal oxytocin: A randomized, placebo-controlled pilot trial. J Psychiatr Res. 2018 Mar;98:64-69. doi: 10.1016/j.jpsychires.2017.12.014. Epub 2017 Dec 26. PMID 29294429

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 8 | 9
Completed | 6 | 7
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.63 (14.58) | 45.78 (15.09) | 43.82 (14.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 3 | 6
  White | 3 | 3 | 6
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptom Severity
Description: Clinician-Administered PTSD Scale (CAPS-5). CAPS-5 scores range from 0-120. Items are summed to obtain a total score with higher scores reflective of greater symptom severity.
Time Frame: Change from Baseline to end of treatment (10 weeks)
Population: Data belonging to participants who completed the trial were examined.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 6 | 7
scores on a scale | 13.00 (12.74) | 17.71 (9.62)

2. Secondary Outcome: PTSD Symptom Severity
Description: PTSD Checklist (PCL). The PCL is a self-report measure which uses a 5-point scale to assess the frequency and severity of PTSD symptoms. Item responses are summed to obtain a total score ranging from 17-85 with greater scores reflective of greater symptom severity.
Time Frame: Change from Baseline to end of treatment (10 weeks)
Population: Data belonging to participants who completed the trial were examined.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 6 | 7
scores on a scale | 20.50 (19.53) | 29.71 (26.39)

3. Secondary Outcome: Depression Symptom Severity
Description: Beck Depression Inventory-II. The BDI-II is a self-report measure where each item is rated on a 0-3 scale and summed to obtain a total score. Greater scores are reflective of greater symptom severity.
Time Frame: Change from Baseline to end of treatment (10 weeks)
Population: Data belonging to participants who completed the trial were examined.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 6 | 7
scores on a scale | 12.67 (11.24) | 17.14 (17.56)

ADVERSE EVENTS:
Time Frame: 2 years.
Description: All adverse events were recorded.
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=8) | Placebo (N=9)
Chest pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No